CLINICAL TRIAL: NCT01900080
Title: Same-Day HIV Testing and Treatment Initiation to Improve Retention in Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic (Other); Weill Medical College of Cornell University (Other); Harvard Medical School (HMS and HSDM) (Other); Florida International University (Other)
Responsible Party: Principal Investigator, Serena Patricia Koenig, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI104344-01A1
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: HIV
Keywords: HIV; AIDS; Antiretroviral therapy; Retention in care; Adherence; Cost-effectiveness
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Same-Day ART Group (Experimental): Same-Day HIV testing and ART initiation:
  All participants in the same-day ART group will receive rapid HIV antibody testing, CD4 cell testing, clinically relevant testing for OIs, WHO staging, counseling and social support, and ART initiation on the day of presentation for HIV testing.
  Interventions: Other: Same-Day HIV testing and ART initiation
- Standard ART Group (Active Comparator): Standard ART Initiation:
  The standard group will receive the same services as the same-day ART group (including same-day HIV and CD4 cell testing) except that instead of same-day ART, they will receive the standard GHESKIO protocol of 3 sequential visits for ART readiness counseling and testing for OIs prior to ART initiation.
  Interventions: Other: Standard ART Initiation
- Sub-Study - Same-Day ART, CD4>500 (Experimental): Sub-Study - Same-Day CD4 Count and ART Initiation for Patients with CD4 Count >500 cells/mm3: Participants will receive counseling and start ART on the day of study enrollment. They will have follow-up visits with the physician on Days 3, 10, 17, and 24, and with the social worker on Days 3, 10, and 17. They will have also have physician visits at weeks 8 and 12. Participants who are clinically stable, asymptomatic, and adherent at week 12 will then qualify for expedited care at future visits, which includes dispensing of ART directly by nurses in the clinic every four weeks, to reduce waiting time for patients. Participants who are symptomatic or non-adherent will be referred to a physician for evaluation.
  Interventions: Other: Sub-Study: Same-Day ART, CD4 Count >500
- Sub-Study - Pre-ART Care, CD4>500 (Active Comparator): Participants will receive standard GHESKIO pre-ART care, which includes a monthly visit with a physician for 3 months, and then every other month physician visits.
  Interventions: Other: Sub-Study: Standard Pre-ART Care, CD4 Count >500

INTERVENTIONS:
Other: Same-Day HIV testing and ART initiation — Same-day HIV testing and ART initiation
  Arms: Same-Day ART Group
Other: Standard ART Initiation — Standard ART Initiation
  Arms: Standard ART Group
Other: Sub-Study: Same-Day ART, CD4 Count >500 — Same-day CD4 count and ART initiation for patients with CD4 count >500 cells/mm3 (CD4 count within 7 days of HIV test)
  Arms: Sub-Study - Same-Day ART, CD4>500
Other: Sub-Study: Standard Pre-ART Care, CD4 Count >500 — Standard pre-ART care for patients with CD4 count >500 cells/mm3
  Arms: Sub-Study - Pre-ART Care, CD4>500

SUMMARY:
The purpose of this study is to determine if same-day HIV testing and antiretroviral therapy (ART) initiation improves retention in care (as measured by the proportion of participants who are alive and in-care with an undetectable viral load 12 months after HIV testing), compared with standard of care (three visits prior to ART initiation). Secondary outcomes include survival, ART initiation, retention in care with viral load < 200 and < 1000 copies/ml, 6-month viral load, and adherence as measured by self-report and pharmacy refill records. Enrollment for the main study was completed in October 2015.

In June 2015, enrollment was started for a new sub-study. This sub-study, funded by MAC AIDS, includes patients with WHO stage 1 or 2 disease and CD4 count >500 cells/mm3. The purpose of the sub-study is to compare 6-month retention for patients who receive same-day ART vs. standard pre-ART care. Secondary outcomes include adherence to INH and Bactrim, and cost-effectiveness between the two groups. Enrollment for the sub-study is ongoing.

DETAILED DESCRIPTION:
This study is a randomized trial to establish the effectiveness of same-day ART initiation for patients who present for HIV testing with early HIV clinical disease (World Health Organization [WHO] stage 1 or 2) who qualify for ART by immunologic criteria (CD4 cell count ≤500 cells/mm3) with rapid CD4 cell testing at the GHESKIO Center in Port-au-Prince, Haiti. All patients in the intervention group received rapid HIV antibody testing, CD4 cell testing, clinically relevant testing for opportunistic infections, WHO staging, comprehensive counseling and social support, and ART initiation on the day of presentation. The standard group received the same services as the same-day ART group (including CD4 cell testing) except that instead of same-day ART, they received the standard GHESKIO protocol of three sequential visits for ART readiness counseling and testing for opportunistic infections prior to ART initiation. For the same-day ART group, these activities took place on the day of ART initiation and during the subsequent two weeks. Three specific aims are proposed. The first aim is to compare the proportion of patients in the standard and same-day ART groups that are alive and in-care with an undetectable HIV viral load at 12 months after HIV testing. The second aim is to compare six-month ART adherence between the two groups using pharmacy refill records. The third aim is to compare the cost and cost-effectiveness of standard and same-day ART, where cost is measured by the mean treatment cost and effectiveness is measured by being alive and in care with an undetectable viral load at 12 months after HIV testing.

In a sub-study funded by MAC AIDS Foundation (enrollment started June 2015), patients with WHO stage 1 or 2 disease and CD4 count >500 cells/mm3 were included. They are being randomized to receive ART vs. standard pre-ART care. Participants are being enrolled in the study on the same day they receive CD4 count results, which is within 7 days of the date of HIV testing. All patients will receive additional tests as clinically indicated. All participants will receive prophylactic treatment with trimethoprim-sulfamethoxazole and isoniazid, and a daily multivitamin, as is standard of care at GHESKIO. Participants who are randomized to the standard pre-ART group will receive standard GHESKIO pre-ART care, which includes a monthly visit with a physician for 3 months, and then every other month physician visits. They will have a CD4 count annually, and start ART when they meet WHO criteria. Participants who are randomized to the same-day ART group will receive counseling and start ART on the day of study enrollment. They will have follow-up visits with the physician on Days 3, 10, 17, and 24, and with the social worker on Days 3, 10, and 17. They will have also have physician visits at weeks 8 and 12. Participants who are clinically stable, asymptomatic, and adherent at week 12 will then qualify for expedited care at future visits, which includes dispensing of ART directly by nurses in the clinic every four weeks, to reduce waiting time for patients. Participants who are symptomatic or non-adherent will be referred to a physician for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Ability and willingness of participant to give written informed consent;
* CD4 cell count </=500 cells/mm3
* WHO stage 1 or 2 disease as defined by the following conditions: Asymptomatic; Persistent generalized lymphadenopathy; Moderate unexplained weight loss (under 10% of presumed or measured body weight); Recurrent upper respiratory tract infections (sinusitis, tonsillitis, otitis media, pharyngitis); Herpes zoster; Angular cheilitis; Recurrent oral ulcerations; Papular pruritic eruptions; Seborrheic dermatitis; Fungal nail infections

Exclusion Criteria:

* Any use of ART in the past;
* Pregnancy or breastfeeding at the screening visit;
* Psychologically unprepared to start ART, based on ART readiness survey;
* Plans to transfer care to another clinic during the study period;
* WHO stage 3 or 4 disease.

Note: For the sub-study that includes patients with WHO stage 1 or 2 disease and CD4 count >500, the inclusion and exclusion criteria are the same; only CD4 count is different.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 814 (Actual)
Dates: Start 2013-08; Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Retention in care with undetectable viral load | 12 months after HIV testing
  Proportion of patients who are alive and in-care with a plasma HIV-1 RNA level <50 copies at 12 months after HIV testing

SECONDARY OUTCOMES:
Adherence to antiretroviral therapy (ART), measured by pharmacy refill records and self-report | 6 months after ART initiation
  Comparison of adherence for the first 6 months of ART between the two groups using pharmacy refill records and 3-day self-report

OTHER OUTCOMES:
Cost-effectiveness | 12 months after HIV testing
  To compare the cost and cost-effectiveness of standard and same-day ART, where cost is measured by the mean treatment cost and effectiveness is measured by being alive and in care with a plasma HIV-1 RNA level <50 copies/ml at 12 months after HIV testing
Retention with undetectable viral load at <200 copies/ml and <1000 copies/ml cut-off points | 6 and 12 months after HIV testing
  Proportion of participants who are alive and in care with a plasma HIV-1 RNA level <200 copies/ml and <1000 copies/ml
ART initiation | 12 months
  Proportion of participants who initiate ART during the study period
Time to Death or LTFU | 12 months
  Median time to death or LTFU

CONTACTS AND LOCATIONS:
Overall Officials: Serena P Koenig, MD, Principal Investigator — Brigham and Women's Hospital; Jean W Pape, MD, Study Director — GHESKIO; Weill Medical College of Cornell University; Marie Marcelle Deschamps, MD, Study Director — Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic
Locations (1):
- Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic Infections (GHESKIO), Port-au-Prince, Haiti

IPD SHARING:
Plan to Share IPD: Yes
Study data will be posted after publication.

REFERENCES:
- [Derived] Koenig SP, Dorvil N, Devieux JG, Hedt-Gauthier BL, Riviere C, Faustin M, Lavoile K, Perodin C, Apollon A, Duverger L, McNairy ML, Hennessey KA, Souroutzidis A, Cremieux PY, Severe P, Pape JW. Same-day HIV testing with initiation of antiretroviral therapy versus standard care for persons living with HIV: A randomized unblinded trial. PLoS Med. 2017 Jul 25;14(7):e1002357. doi: 10.1371/journal.pmed.1002357. eCollection 2017 Jul. PMID 28742880